CLINICAL TRIAL: NCT02663648
Title: Cell Cycle Regulatory Gene Study in Patients With Myeloproliferative Disorders
Status: Withdrawn | Type: Observational
Why Stopped: No eligible patient was enrolled.
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Other Study IDs: Cell cycle regulatory gene-MPD
Record Dates: First submitted 2015-12-21; First posted 2016-01-26 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-01

CONDITIONS: Myeloproliferative Disorders; Polycythemia Vera; Essential Thrombocythemia; Myelofibrosis; Chronic Myeloid Leukemia
Keywords: myeloproliferative disorders; cell cycle regulatory protein
MeSH Terms: conditions — Myeloproliferative Disorders; Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study involves observing the level of cell cycle regulatory gene in patients with myeloproliferative disorders(MPD). These disorders include polycythemia vera (PV), essential thrombocythemia (ET), myelofibrosis (MF) and chronic myeloid leukemia (CML). The abnormal blood and/or bone marrow cells, or materials derived from these abnormal cells, like DNA, RNA, protein or plasma will be used in laboratory studies.

Cell cycle regulatory protein such as cyclins, cyclin-dependent kinases(Cdks) and Cdk inhibitors(CKIs) play indispensable roles in processes such as transcription, metabolism and stem cell self-renewal. MPD are a group of diseases characterized by abnormally increased proliferation of erythroid, megakaryocytic, or granulocytic cells. The pathogenesis was still unclear. Detecting the level of cell cycle regulatory protein will be useful to look for the possible role in MPD and better understand the cause of MPD.

DETAILED DESCRIPTION:
This study involves observing the level of cell cycle regulatory gene in patients with myeloproliferative disorders(MPD). These disorders include polycythemia vera (PV), essential thrombocythemia (ET), myelofibrosis (MF) and chronic myeloid leukemia (CML). The abnormal blood and/or bone marrow cells, or materials derived from these abnormal cells, like DNA, RNA, protein or plasma will be used in laboratory studies.

Cell cycle regulatory protein such as cyclins, cyclin-dependent kinases(Cdks) and Cdk inhibitors(CKIs) play indispensable roles in processes such as transcription, metabolism and stem cell self-renewal. MPD are a group of diseases characterized by abnormally increased proliferation of erythroid, megakaryocytic, or granulocytic cells. The pathogenesis was still unclear. Detecting the level of cell cycle regulatory protein will be useful to look for the possible role in MPD and better understand the cause of MPD.

In this study, the cell cycle regulatory message RNA and protein from patients' and healthy volunteers' bone marrow and peripheral blood will be extracted and quantified by real time polymerase chain reaction and western blot. The different level of cell cycle regulatory gene between patients and volunteers and the relationship between the level and patients' clinical characteristics such as age, gender, type of disease will be analysed by SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of polycythemia vera (PV), essential thrombocythemia (ET), myelofibrosis (MF) or chronic myeloid leukemia (CML) as defined by the World Health Organization (WHO) diagnostic criteria

Exclusion Criteria:

* Have received treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Have a diagnosis of polycythemia vera (PV), essential thrombocythemia (ET), myelofibrosis (MF) or chronic myeloid leukemia (CML) as defined by the World Health Organization (WHO) diagnostic criteria
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
quantified the level of CDK, CCP, PLK by real time PCR and westen blot | two years
  The cell cycle regulatory message RNA and protein from patients' and healthy volunteers' bone marrow and peripheral blood will be extracted and quantified by real time polymerase chain reaction and western blot. The cell cycle regulatory genes contain CDK ,CDKI, Ser/Thr protein kinase, ATP/GTP binding protein-like and so on.
age of MPN patients and volunteers | two years
  observe the age of MPN patients and volunteers, and analyze the correlation between the level and the age of patients.
gender of MPN patients and volunteers | two years
  observe different level of cell cycle regulatory gene between male patients and femal patients.
count of peripheral blood cells | two years
  observe the count of peripheral blood cells, including the white blood cell, red blood cell and platelet.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Peng, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China